CLINICAL TRIAL: NCT03914989
Title: Sensory Enrichment for Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to complete full enrollment due to Covid pandemic.
Sponsor: University of California, Irvine (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Principal Investigator, Michael Leon, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014-1078
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-02

CONDITIONS: Cognitive Function
Keywords: Memory preservation; Age-related memory disorders; Intervention; Life quality; Olfaction
MeSH Terms: conditions — Memory Disorders; Anosmia | interventions — Oils, Volatile

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an experimental group or an active control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the participants and the assessors will be blinded to the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Individuals in this group receive exposure to a higher concentration of essential oil fragrances nightly.
  Interventions: Other: olfactory enrichment (essential oils)
- Active control group (Placebo Comparator): Individuals in this group receive exposure to a lower concentration of essential oil fragrances nightly.
  Interventions: Other: olfactory enrichment (essential oils)

INTERVENTIONS:
Other: olfactory enrichment (essential oils) — Participants will be exposed to either a higher or lower concentration of essential oils nightly for two hours as they are going to sleep, using a nebulizing fragrance diffuser, rotating through seven different scents, one per night.

SUMMARY:
This study evaluates the efficacy of multi-odorant enrichment on cognitive skills, olfactory function, and quality of life.

DETAILED DESCRIPTION:
The purpose of this study is to explore sensory stimulation as a potential means of enhancing cognitive abilities. In mice, multi-odorant enrichment has been shown to increase neurogenesis in a critical memory pathway and thereby improve memory. In this clinical study, we will determine if a nightly sensory enrichment regimen using scents for 6 months can improve cognitive skills, as measured using a series of cognitive assessments and brain imaging in older adults. We also will determine if mood/mental state of mind or olfactory functioning improve following scent stimulation.

This study will enroll approximately 200 participants. Of the 200 participants in the study, 50 individuals, who are interested in participating, will have a functional Magnetic Resonance Imaging (fMRI) scan at the beginning and end of the study, which will be used to examine changes in the brain.

Participants will undergo cognitive assessments, computerized cognitive assessments, and olfactory function assessments. They will be randomly assigned to either an experimental or an active control group, and will be exposed to either a higher or lower concentration of essential oils nightly using a nebulizing fragrance diffuser, rotating through seven different scents, one per night. The exposures will continue for 6 months, after which the participants will return and undergo the same assessments conducted at the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Are age 60-85, male or female
2. Have normal cognition (determined at first assessment with cognitive testing)
3. Speak/read/understand English fluently
4. Have visual and auditory acuity adequate for neuropsychological and computerized testing
5. Are in good general health with no disease(s) expected to interfere with the study
6. Are willing and able to participate for the duration of the study and in all study procedures
7. Are able to smell scents
8. Are willing to refrain from using scented candles, scented oils, or air fresheners while participating in the study
9. Are willing to travel to the research site for testing

   If interested in functional Magnetic Resonance Imaging (fMRI),
10. Are willing and able to participate in the fMRI scan.

Exclusion Criteria:

1. Have known fragrance sensitivities
2. Have asthma, allergies, or a fragrance sensitivity, which produces symptoms similar to those of an allergy, including runny nose, watery eyes, sneezing, or skin rash
3. Have a neurologic disease such as Parkinson's disease, multiple sclerosis, brain cyst, tumor or aneurysm
4. Have major health conditions such as uncontrolled diabetes mellitus, uncontrolled hypertension, nutritional deficiency or thyroid disease
5. Have significant psychiatric disorders such as schizophrenia, bipolar disorder, anxiety disorder, or attention-deficit hyperactivity disorder
6. Have cognitive impairment when tested at baseline (defined as a score on any neuropsychological test of 1.5 standard deviations or more outside the age norm)
7. Have had alcohol or substance abuse or dependence within the past 2 years (DSM-IV criteria)
8. Smoke cigarettes, e-cigarettes, cigars, marijuana, or any other substance that could produce an interfering odor for the study.

   If interested in functional Magnetic Resonance Imaging (fMRI),
9. MRI contraindications, (e.g. pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of behavioral pattern separation ability | 1) at Baseline and 2) after 6 months of intervention
  Change in lure discrimination index on a computerized mnemonic discrimination task.

SECONDARY OUTCOMES:
Evaluation of cognition | 1) at Baseline and 2) after 6 months of intervention
  Change in cognitive ability will be measured using scores from a neuropsychological battery. For each subsection, a change score will be calculated using the difference between baseline and 6-month scores, and the change score will be compared between groups. Higher values indicate a better outcome.
Evaluation of depression | 1) at Baseline and 2) after 6 months of intervention
  Change in depression status using the Beck Depression Inventory.
Evaluation of quality of life | 1) at Baseline and 2) after 6 months of intervention
  Change in quality of life using the Farage Quality of Life questionnaire.
Evaluation of olfactory function | 1) at Baseline and 2) after 6 months of intervention
  Change from baseline score on the Sniffin' Sticks instrument to assess olfactory system functioning.
Evaluation of change in brain structural connectivity | 1) at Baseline and 2) after 6 months of intervention
  Change in perforant path integrity using functional Magnetic Resonance Imaging.
Evaluation of change in brain structures | 1) at Baseline and 2) after 6 months of intervention
  Change in thickness of entorhinal cortex using functional Magnetic Resonance Imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Leon, PhD, Principal Investigator — University of California, Irvine; Michael Yassa, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No